CLINICAL TRIAL: NCT03346525
Title: The GOAL (GwokO Adunu pa Lutino) Trial: Determining the Impact of Penicillin on Latent Rheumatic Heart Disease: A Randomized Controlled Trial in Uganda
Brief Title: Determining the Impact of Penicillin in Latent RHD: The GOAL Trial
Acronym: GOAL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Children's National Research Institute (Other)
Collaborators: Thrasher Research Fund (Other); University of Cape Town (Other); Uganda Heart Institute (Other); Karp Family Foundation (Unknown); Gift of Life International (Other); Murdoch Childrens Research Institute (Other)
Responsible Party: Principal Investigator, Andrea Beaton, Pediatric Cardiologist, Associate Professor of Pediatrics, Children's Hospital Medical Center, Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GOAL: RHD RCT; E.W. "Al" Thrasher Award (Other: Thrasher Research Fund)
Record Dates: First submitted 2017-11-15; First posted 2017-11-17 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Rheumatic Heart Disease in Children; Latent Rheumatic Heart Disease; Rheumatic Heart Disease; Heart Diseases
Keywords: echocardiography; penicillin prophylaxis; intramuscular benzathine penicillin G; benzathine penicillin G; low-resource setting
MeSH Terms: conditions — Rheumatic Heart Disease; Heart Diseases | interventions — Penicillin G

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BPG Arm (Experimental): Intramuscular BPG prophylaxis (600,000 IU for children <30kg, 1.2 million IU for children ≥30kg), every 28 days
  Interventions: Drug: intramuscular benzathine penicillin G (BPG) prophylaxis
- Control Arm (No Intervention): No prophylaxis

INTERVENTIONS:
Drug: intramuscular benzathine penicillin G (BPG) prophylaxis — Intramuscular BPG prophylaxis (600,000 IU for children <30kg, 1.2 million IU for children ≥30kg), every 28 days.
  Other Names: benzathine penicillin G; BPG; penicillin prophylaxis
  Arms: BPG Arm

SUMMARY:
Rheumatic heart disease (RHD) affects at least 32.9 million people, mostly children living in low-resource settings. Long-term intramuscular benzathine penicillin G (BPG) prophylaxis is proven to prevent progression of chronic valve changes in patients with established rheumatic heart disease (RHD) and to allow regression of valve changes in patients with a history of acute rheumatic fever (ARF) with mild RHD. However, in low-resource settings ARF is an elusive diagnosis, and most patients (85%) are diagnosed only when RHD is severe and irreversible, medications ineffective, and surgical intervention is expensive and/or unavailable.

Identification of latent RHD might be an opportunity to substantially reduce RHD morbidity and mortality. However, detection of latent RHD is only important if outcomes are improved. The appropriate management of children with latent RHD is unknown and no formal recommendations exist. While some clinicians prescribe penicillin prophylaxis for children with latent RHD, clinical equipoise exists regarding the best practice.

To fill this gap, the investigators propose a randomized controlled trial in children with latent RHD to evaluate the efficacy of BPG prophylaxis compared to no prophylaxis. Our primary outcome measure is progression of valvular changes on echocardiogram at 2 years. A sample size of 916 children is needed to detect a 50% reduction of progression (expected range 7.5-12.5% progression in BPG-arm vs. 15%-25% progression in control-arm) with 90% power.

AIM 1: To compare the proportion of children (aged 5-17 years) with latent RHD receiving BPG prophylaxis who progress to worse valvular disease at 2-years compared to children not receiving BPG prophylaxis.

Hypothesis 1: Prophylaxis with BPG will result in fewer children with latent RHD showing progression of echocardiographic valve changes at 2 years compared to children with latent RHD not receiving BPG prophylaxis. (The investigators expect at least a 50% relative reduction in progression in the BPG arm: range 15%-25% control arm vs. 7.5-12.5% BPG-arm.)

AIM 2: To compare the proportion of children (aged 5-17 years) with latent RHD receiving BPG prophylaxis who regress to improved valvular disease at 2-years compared to children not receiving BPG prophylaxis.

Hypothesis 2: Prophylaxis with BPG will result in more children with latent RHD showing regression of echocardiographic valve changes by 2 years compared to children with latent RHD not receiving BPG prophylaxis. (The investigators expect at least a 50% relative increase in regression in the BPG arm: range 10-20% control arm vs. 20-40% BPG arm.)

This study is highly significant because it will establish if BPG prophylaxis improves outcomes for children with latent RHD. Feasibility will be ensured through the experience, resources, community support, and accessible patient population of our investigational team. The results of our study will have high impact, immediately informing international policy on the standard of care for children diagnosed with latent RHD and shaping, over 2-3 years, practical and scalable programs that could substantially decrease the global burden of RHD.

ELIGIBILITY:
Inclusion Criteria:

* Children will be eligible for study participation if they are (1) between the ages of 5-17 years and (2) have a new diagnosis of latent RHD detected through primary school echo screening and confirmed by blinded consensus review. All children will be recruited from schools in Gulu District in Uganda.

Exclusion Criteria:

* Patients will be excluded from the study for the following reasons:

  * Known history of ARF or RHD
  * Newly diagnosed RHD by echo screening consider to be "missed clinical RHD" as compared to true latent RHD including: > mild pathological valvular regurgitation at the mitral valve or aortic valve, mitral stenosis (mean MV gradient ≥ 5mmHg) (WHF, definite B), aortic stenosis (mean AV gradient ≥ 20mmHg)
  * Structural or functional cardiac defects, other than those consistent with RHD, that were known prior to or detected through echo screening (except patent foramen ovale, small atrial septal defect, small ventricular septal defect, small patent ductus arteriosus).
  * Prior allergic reaction to penicillin
  * Any known conditions predisposing to thrombocytopenia or hypercoagulability, or other contraindications to intramuscular injection
  * Any known co-morbid conditions (HIV, renal deficiencies, severe malnutrition among others) that have resulted in prescription of regular antibiotic prophylaxis

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 807 (Actual)
Dates: Start 2018-06-26 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
progression of valvular changes on echocardiogram at 2 years | 2 years
  To compare the proportion of children (aged 5-17 years) with latent RHD receiving BPG prophylaxis who progress to worse valvular disease at 2-years compared to children not receiving BPG prophylaxis

SECONDARY OUTCOMES:
regression of vavular changes on electrocardiogram at 2 years | 2 years
  To compare the proportion of children (aged 5-17 years) with latent RHD receiving BPG prophylaxis who regress to improved valvular disease at 2-years compared to children not receiving BPG prophylaxis

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Beaton, MD, Principal Investigator — Cincinnati Children's
Locations (1):
- GOAL Office, Gulu, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] WHO - Global Burden of Disease. 2015;2015.
- [Background] Lue HC, Wu MH, Wang JK, Wu FF, Wu YN. Long-term outcome of patients with rheumatic fever receiving benzathine penicillin G prophylaxis every three weeks versus every four weeks. J Pediatr. 1994 Nov;125(5 Pt 1):812-6. doi: 10.1016/s0022-3476(94)70082-6. PMID 7965439
- [Background] Tompkins DG, Boxerbaum B, Liebman J. Long-term prognosis of rheumatic fever patients receiving regular intramuscular benzathine penicillin. Circulation. 1972 Mar;45(3):543-51. doi: 10.1161/01.cir.45.3.543. No abstract available. PMID 5012243
- [Background] Zhang W, Mondo C, Okello E, Musoke C, Kakande B, Nyakoojo W, Kayima J, Freers J. Presenting features of newly diagnosed rheumatic heart disease patients in Mulago Hospital: a pilot study. Cardiovasc J Afr. 2013 Mar;24(2):28-33. doi: 10.5830/CVJA-2012-076. PMID 23612950
- [Background] Okello E, Wanzhu Z, Musoke C, Twalib A, Kakande B, Lwabi P, Wilson NB, Mondo CK, Odoi-Adome R, Freers J. Cardiovascular complications in newly diagnosed rheumatic heart disease patients at Mulago Hospital, Uganda. Cardiovasc J Afr. 2013 Apr;24(3):80-5. doi: 10.5830/CVJA-2013-004. PMID 23736132
- [Background] Beaton A, Okello E, Lwabi P, Mondo C, McCarter R, Sable C. Echocardiography screening for rheumatic heart disease in Ugandan schoolchildren. Circulation. 2012 Jun 26;125(25):3127-32. doi: 10.1161/CIRCULATIONAHA.112.092312. Epub 2012 May 24. PMID 22626741
- [Background] Steer AC, Kado J, Wilson N, Tuiketei T, Batzloff M, Waqatakirewa L, Mulholland EK, Carapetis JR. High prevalence of rheumatic heart disease by clinical and echocardiographic screening among children in Fiji. J Heart Valve Dis. 2009 May;18(3):327-35; discussion 336. PMID 19557993
- [Background] Engel ME, Haileamlak A, Zuhlke L, Lemmer CE, Nkepu S, van de Wall M, Daniel W, Shung King M, Mayosi BM. Prevalence of rheumatic heart disease in 4720 asymptomatic scholars from South Africa and Ethiopia. Heart. 2015 Sep;101(17):1389-94. doi: 10.1136/heartjnl-2015-307444. Epub 2015 Jun 15. PMID 26076935
- [Background] Zuhlke LJ, Beaton A, Engel ME, Hugo-Hamman CT, Karthikeyan G, Katzenellenbogen JM, Ntusi N, Ralph AP, Saxena A, Smeesters PR, Watkins D, Zilla P, Carapetis J. Group A Streptococcus, Acute Rheumatic Fever and Rheumatic Heart Disease: Epidemiology and Clinical Considerations. Curr Treat Options Cardiovasc Med. 2017 Feb;19(2):15. doi: 10.1007/s11936-017-0513-y. PMID 28285457
- [Background] Remenyi B, Wilson N, Steer A, Ferreira B, Kado J, Kumar K, Lawrenson J, Maguire G, Marijon E, Mirabel M, Mocumbi AO, Mota C, Paar J, Saxena A, Scheel J, Stirling J, Viali S, Balekundri VI, Wheaton G, Zuhlke L, Carapetis J. World Heart Federation criteria for echocardiographic diagnosis of rheumatic heart disease--an evidence-based guideline. Nat Rev Cardiol. 2012 Feb 28;9(5):297-309. doi: 10.1038/nrcardio.2012.7. PMID 22371105
- [Background] Beaton A, Lu JC, Aliku T, Dean P, Gaur L, Weinberg J, Godown J, Lwabi P, Mirembe G, Okello E, Reese A, Shrestha-Astudillo A, Bradley-Hewitt T, Scheel J, Webb C, McCarter R, Ensing G, Sable C. The utility of handheld echocardiography for early rheumatic heart disease diagnosis: a field study. Eur Heart J Cardiovasc Imaging. 2015 May;16(5):475-82. doi: 10.1093/ehjci/jeu296. Epub 2015 Jan 5. PMID 25564396
- [Background] Weinberg J, Beaton A, Aliku T, Lwabi P, Sable C. Prevalence of rheumatic heart disease in African school-aged population: Extrapolation from echocardiography screening using the 2012 World Heart Federation Guidelines. Int J Cardiol. 2016 Jan 1;202:238-9. doi: 10.1016/j.ijcard.2015.08.128. Epub 2015 Sep 12. No abstract available. PMID 26402451
- [Background] Roberts K, Colquhoun S, Steer A, Remenyi B, Carapetis J. Screening for rheumatic heart disease: current approaches and controversies. Nat Rev Cardiol. 2013 Jan;10(1):49-58. doi: 10.1038/nrcardio.2012.157. Epub 2012 Nov 13. PMID 23149830
- [Background] Karthikeyan G. Measuring and reporting disease progression in subclinical rheumatic heart disease. Heart Asia. 2016 Nov 28;8(2):74-75. doi: 10.1136/heartasia-2016-010857. eCollection 2016. No abstract available. PMID 27942046
- [Background] Nascimento BR, Nunes MC, Lopes EL, Rezende VM, Landay T, Ribeiro AL, Sable C, Beaton AZ. Rheumatic heart disease echocardiographic screening: approaching practical and affordable solutions. Heart. 2016 May;102(9):658-64. doi: 10.1136/heartjnl-2015-308635. Epub 2016 Feb 18. PMID 26891757
- [Background] Steer AC, Romani L, Kaldor JM. Mass Drug Administration for Scabies Control. N Engl J Med. 2016 Apr 28;374(17):1690. doi: 10.1056/NEJMc1600495. No abstract available. PMID 27119244
- [Background] Engelman D, Okello E, Beaton A, Selnow G, Remenyi B, Watson C, Longenecker CT, Sable C, Steer AC. Evaluation of Computer-Based Training for Health Workers in Echocardiography for RHD. Glob Heart. 2017 Mar;12(1):17-23.e8. doi: 10.1016/j.gheart.2015.12.001. Epub 2016 Mar 16. PMID 26994642
- [Background] Ploutz M, Lu JC, Scheel J, Webb C, Ensing GJ, Aliku T, Lwabi P, Sable C, Beaton A. Handheld echocardiographic screening for rheumatic heart disease by non-experts. Heart. 2016 Jan;102(1):35-9. doi: 10.1136/heartjnl-2015-308236. Epub 2015 Oct 5. PMID 26438784
- [Background] Lopes EL, Beaton AZ, Nascimento BR, Tompsett A, Dos Santos JP, Perlman L, Diamantino AC, Oliveira KK, Oliveira CM, Nunes MDCP, Bonisson L, Ribeiro AL, Sable C; Programa de RastreamentO da Valvopatia Reumatica (PROVAR) investigators. Telehealth solutions to enable global collaboration in rheumatic heart disease screening. J Telemed Telecare. 2018 Feb;24(2):101-109. doi: 10.1177/1357633X16677902. Epub 2016 Nov 4. PMID 27815494
- [Background] Zhang W, Okello E, Nyakoojo W, Lwabi P, Mondo CK. Proportion of patients in the Uganda rheumatic heart disease registry with advanced disease requiring urgent surgical interventions. Afr Health Sci. 2015 Dec;15(4):1182-8. doi: 10.4314/ahs.v15i4.17. PMID 26958019
- [Background] Okello E, Longenecker CT, Beaton A, Kamya MR, Lwabi P. Rheumatic heart disease in Uganda: predictors of morbidity and mortality one year after presentation. BMC Cardiovasc Disord. 2017 Jan 7;17(1):20. doi: 10.1186/s12872-016-0451-8. PMID 28061759
- [Background] Beaton A, Okello E, Aliku T, Lubega S, Lwabi P, Mondo C, McCarter R, Sable C. Latent rheumatic heart disease: outcomes 2 years after echocardiographic detection. Pediatr Cardiol. 2014 Oct;35(7):1259-67. doi: 10.1007/s00246-014-0925-3. Epub 2014 May 15. PMID 24827080
- [Derived] Beaton A, Okello E, Rwebembera J, Grobler A, Engelman D, Alepere J, Carapetis J, DeWyer A, Lwabi P, Mirabel M, Mocumbi AO, Nakitto M, Ndagire E, Nunes MCP, Omara IO, Sarnacki R, Scheel A, Wilson N, Zuhlke L, Karthikeyan G, Sable CA, Steer AC. Refining Risk Stratification Among Children With Latent Rheumatic Heart Disease. Circulation. 2023 Jun 13;147(24):1848-1850. doi: 10.1161/CIRCULATIONAHA.122.063194. Epub 2023 Jun 12. No abstract available. PMID 37307310
- [Derived] Beaton A, Okello E, Rwebembera J, Grobler A, Engelman D, Alepere J, Canales L, Carapetis J, DeWyer A, Lwabi P, Mirabel M, Mocumbi AO, Murali M, Nakitto M, Ndagire E, Nunes MCP, Omara IO, Sarnacki R, Scheel A, Wilson N, Zimmerman M, Zuhlke L, Karthikeyan G, Sable CA, Steer AC. Secondary Antibiotic Prophylaxis for Latent Rheumatic Heart Disease. N Engl J Med. 2022 Jan 20;386(3):230-240. doi: 10.1056/NEJMoa2102074. Epub 2021 Nov 13. PMID 34767321
- [Derived] Scheel A, Mirabel M, Nunes MCP, Okello E, Sarnacki R, Steer AC, Engelman D, Zimmerman M, Zuhlke L, Sable C, Beaton A. The inter-rater reliability and individual reviewer performance of the 2012 world heart federation guidelines for the echocardiographic diagnosis of latent rheumatic heart disease. Int J Cardiol. 2021 Apr 1;328:146-151. doi: 10.1016/j.ijcard.2020.11.013. Epub 2020 Nov 10. PMID 33186665
- [Derived] Beaton A, Okello E, Engelman D, Grobler A, Scheel A, DeWyer A, Sarnacki R, Omara IO, Rwebembera J, Sable C, Steer A. Determining the impact of Benzathine penicillin G prophylaxis in children with latent rheumatic heart disease (GOAL trial): Study protocol for a randomized controlled trial. Am Heart J. 2019 Sep;215:95-105. doi: 10.1016/j.ahj.2019.06.001. Epub 2019 Jun 8. PMID 31301533